CLINICAL TRIAL: NCT00673543
Title: The Effects of Corticosteroid Therapy on Glucose Control in Pregnant Women With Insulin Requiring Diabetes Mellitus
Brief Title: Corticosteroid Therapy on Glucose Control in Pregnant Women With Diabetes
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jerrie Refuerzo, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-08-0074
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Pregnant Women
Keywords: Corticosteroids; Pregnancy; Glucose control

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Pregnant women with insulin requiring diabetes
- 2: Pregnant women without insulin requiring diabetes

SUMMARY:
Preterm birth occurs in 25% of women with insulin requiring diabetes in pregnancy. The administration of corticosteroid therapy to accelerate fetal lung maturation is indicated in women at risk for preterm birth. The purpose of this study is to compare the timing, duration and severity of maternal hyperglycemia after corticosteroid administration in women with insulin-requiring diabetes compared to those without diabetes in pregnancy.

This is a prospective, observational study. Hourly glucose levels will be obtained for a total of 7 days after corticosteroid administration using the Dexcom Seven continuous glucose monitoring system. In addition, hemoglobin A1C will be obtained to assess the overall level of glycemic control of the participant prior to the corticosteroid therapy.

DETAILED DESCRIPTION:
Preterm birth occurs in 25% of women with insulin requiring diabetes in pregnancy. The administration of corticosteroid therapy to accelerate fetal lung maturation is indicated in women at risk for preterm birth. Although corticosteroid therapy significantly decreases the risk for respiratory distress syndrome in the newborn, such therapy can lead to transient elevations in maternal glucose levels, potentially resulting in life-threatening maternal metabolic abnormalities, low oxygen levels in the fetus, and in extreme cases, stillbirth. Because the elevations in glucose levels may drastically increase over a short period of time, intense monitoring of maternal glucose levels to achieve strict glycemic control and treatment is preferred with the use of insulin. The purpose of this study is to compare the timing, duration and severity of maternal hyperglycemia after corticosteroid administration in women with insulin-requiring diabetes compared to those without diabetes in pregnancy.

This is a prospective, observational study. Hourly glucose levels will be obtained for a total of 7 days after corticosteroid administration using the Dexcom Seven continuous glucose monitoring system. In addition, hemoglobin A1C will be obtained to assess the overall level of glycemic control of the participant prior to the corticosteroid therapy.

The study group will include pregnant women > 18 years of age with insulin-requiring diabetes who will receive corticosteroid therapy to accelerate fetal lung maturation between 24 and 34 weeks of pregnancy. Only those women not in active labor and with singleton gestations will be included. A control group will be comprised of pregnant women with singleton gestations without insulin-requiring diabetes who will receive corticosteroid therapy also to accelerate fetal lung maturation.

Women will be excluded if they have diet controlled diabetes, twins or higher gestation, are in active labor and anticipate imminent delivery, were previously on any form of steroid therapy, or who have or will be receiving beta-adrenergic medications.

ELIGIBILITY:
Inclusion Criteria:

* The study group will include pregnant women > 18 years of age with insulin-requiring diabetes who will receive corticosteroid therapy to accelerate fetal lung maturation between 24 and 34 weeks of pregnancy. Only those women not in active labor and with singleton gestations will be included. A control group will be comprised of pregnant women with singleton gestations without insulin-requiring diabetes who will receive corticosteroid therapy also to accelerate fetal lung maturation.

Exclusion Criteria:

* Women will be excluded if they have diet controlled diabetes, twins or higher gestation, are in active labor and anticipate imminent delivery, were previously on any form of steroid therapy, or who have or will be receiving beta-adrenergic medications.

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women who will receive corticosteroid therapy.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2008-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Time point at which glucose elevation occurs after glucocorticoid administration (greater than 50% increase in the patient's baseline blood) glucose level. | Within 7 days

SECONDARY OUTCOMES:
Time at which glucose normalization occurs (ability to achieve glucose level within 20% of the patient's baseline blood glucose level) | 7 days
The change in glucose in incremental amounts (every 4, 6, and 8 hour intervals) over time. | 7 days
The amount of insulin needed to achieve targeted glucose levels over time | 7 days
Total amount of insulin as well as incremental amounts of insulin every (4, 6, and 8 hour intervals) | 7 days
Maternal age | 7 days
Maternal body mass index | 7 days
Gestational age | 7 days
Hemoglobin A1C | 7 days
Pre-corticosteroid insulin amount | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jerrie S Refuerzo, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Lyndon B. Johnson Hospital, Houston, Texas
  - Memorial Hermann Hospital Texas Medical Center, Houston, Texas